CLINICAL TRIAL: NCT03235999
Title: The Experiences of Patients Living With Malignant Pleural Effusions
Status: Completed | Type: Observational
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 16/009/GHT
Record Dates: First submitted 2017-04-12; First posted 2017-08-01 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Talc pleurodesis: Up to 10 patients who have had talc pleurodesis
- IPC: Up to 10 patients who have had indwelling pleural catheters (IPC)

SUMMARY:
Up to 20 patients with malignant pleural effusions will be interviewed about their experiences of having this condition and its management.

ELIGIBILITY:
Inclusion Criteria:

1. Adults diagnosed with a malignant pleural effusion
2. Has undergone either talc pleurodesis or IPC
3. Have signed a consent form prior to entering the study
4. Life expectancy > 6 weeks based on LENT guidelines (Low/Moderate risk group) - The LENT score calculation assigns 0 (<1500 IU/L) or 1 (>1500 IU/L) for pleural fluid LDH level; 0 to 3 points for matching ECOG performance scores (3 and 4 are combined); 0 (<9) or 1 (>9) for neutrophil-to-lymphocyte ratio; and 0 (lowest risk), 1 (moderate risk), or 3 (highest risk) for tumor type.

Exclusion Criteria:

1. Any patient who is unable to understand sufficient English to take part in the semi-structured interviews
2. Weakness or fatigue sufficient so that the patient is unable to take part in the interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant pleural effusions
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Patient Experiences of living with malignant pleural effusion and different pleural procedures | 4 weeks after IPC placement or talc pleurodesis
  Qualitative interviews - Interviews will be recorded on a digital audio recorder and then downloaded on to a password protected computer. The interviews will then be sent for transcription using secure email and anonymised.
  We will perform thematic analysis on the interview data. This is a process to help explore the experiences of the subject as they describe it rather than looking at how they talk about the experience. Themes will be drawn from the data following coding. Common codes relating to a theme, for example pain, will be identified and examples of text used to demonstrate the theme extracted. This will ensure a wide variety of quotes across the interviews rather than focusing on one main or a subset of interviews. We will use an inductive approach whereby themes will emerge and not be developed in advance. Emerging codes will be checked by the supervisory team.
  There will be no numerical, quantitative data for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Perkins, MBBCh, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust
Locations (1):
- Gloucestershire Hospitals NHS Foundation Trust, Cheltenham, Gloucestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No